CLINICAL TRIAL: NCT01559610
Title: Preoperatively Orientation in Cardiac Surgery: Nurses Intervention on Patients Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UP 4150/08
Record Dates: First submitted 2012-02-23; First posted 2012-03-21 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Artery Bypass Graft Triple Vessel; Heart Valve Diseases
Keywords: cardiac surgery; orientation; nursing
MeSH Terms: conditions — Heart Valve Diseases; Orientation, Spatial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Received preoperative guidance by a member of healthcare team with the aid of checklist
  Interventions: Other: Intervention Group
- Group intervention (Other): preoperative guideline by a nurse
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Intervention Group — The patients were instructed by a nurse
  Other Names: No applicable

SUMMARY:
The purpose of this study is to determine whether the guidelines preoperative performed by a nurse contribute to the recovery of the patient submitted to cardiac surgery compared with the guidelines for routine.

DETAILED DESCRIPTION:
This is a randomized clinical trial, which included patients submitted to cardiac surgery on both sexes. They are divided in two groups: control group and intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Primary Elective Cardiac Surgical Procedures
* Age above 18 years old
* At least 24 hours of hospitalization before the procedure

Exclusion Criteria:

* Patients who do not accept and do not signed a consenting term

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
knowledge | seven days
  three questions applied on the second day of recovery at the nursery room, after the intensive care unit discharge,about type of anesthesia,endotracheal tube function and time of healing of the sternum bone.The questions had only one correct alternative.Since the randomization until the questionnaire,the study follow up took seven days.For the analysis,answers of the questionnaire were separated and the number of answers for each,and divided into the two groups.The results were presented in graphic and tables.

SECONDARY OUTCOMES:
satisfaction | seven days
  five questions applied on the second day of recovery at the nursery room.The patients had to graduate their level of satisfaction from unsatisfied to very satisfied according to orientation received about the prior,intraoperative and recovering period of surgery as well as the nursery and medical orientation provided.Since the randomization until the questionnaire,the study follow up took seven days.For the analysis answers of the questionnaire were separated and the number of answers for each,and divided into the two groups.The results were presented in graphic and tables.

CONTACTS AND LOCATIONS:
Overall Officials: Juliane A Rodrigues, nursing, Principal Investigator — Brasil:Instituto de Cardiologia do Rio Grande do Sul/Fundacao Universitaria de Cardiologia
Locations (1):
- Institute of Cardiology, Porto Alegre, Rio Grande do Sul, Brazil